CLINICAL TRIAL: NCT05543681
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Trial of the Safety and Efficacy of IGC-AD1 on Agitation in Participants With Dementia Due to Alzheimer's Disease
Brief Title: Clinical Trial on Agitation in Alzheimer's Dementia
Acronym: CALMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IGC Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IGC-AD1-P2 BIDAG
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Agitation,Psychomotor; Care Giving Burden; NPS; Aggression
Keywords: Cannabis; Tetrahydrocannabinol; THC; Melatonin; Alzheimer's; Marijuana; Hemp; Agitation; Dementia; Depression; Anxiety; NPI; CMAI; Dronabinol
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Caregiver Burden; Aggression; Marijuana Abuse; Dementia; Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multi-site, Randomized, double-blind, placebo-controlled parallel-group trial in adults with mild to severe dementia from Alzheimer's and symptomatological Agitation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind for study site and participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Comparator: IGC-AD1Active (Active Comparator): IGC-AD1-Active, oral solution with two APIs (THC and melatonin).
  Interventions: Drug: IGC-AD1-Active
- Placebo Comparator: IGC-AD1 Placebo (Placebo Comparator): IGC-AD1-Placebo, oral solution similar to Active in color, taste, and texture, with excipients but without APIs.
  Interventions: Drug: IGC-AD1-Placebo

INTERVENTIONS:
Drug: IGC-AD1-Active — A non-sterile solution for oral administration.
  Other Names: Active
  Arms: Active Comparator: IGC-AD1Active
Drug: IGC-AD1-Placebo — A non-sterile solution for oral administration similar in color and texture to the Active.
  Other Names: Placebo
  Arms: Placebo Comparator: IGC-AD1 Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of the oral medication IGC-AD1, a THC-based (Delta-9-Tetrahydrocannabinol) formulation administered twice a day on Agitation in patients with mild to severe dementia from Alzheimer's.

DETAILED DESCRIPTION:
CALMA is a multi-center, double-blind, randomized, placebo-controlled clinical trial. The study targets participants aged 60 and older with mild to severe Alzheimer's dementia who have exhibited clinically significant agitation for at least two weeks prior to enrollment. Agitation caused by other conditions or transient symptoms must be ruled out. Eligibility is determined by a baseline Neuropsychiatric Inventory (NPI-12), Agitation subscale score of ≥4 and the International Psychogeriatric Association (IPA) criteria for agitation.

The investigational medication is an oral solution containing two active ingredients: delta-9 tetrahydrocannabinol (THC) and melatonin. The treatment is administered for 42 days, followed by a two-day taper period at the end of the study.

Safety oversight includes daily calls on days 2, 3, and 4, transitioning to calls every third day thereafter. These calls will review study partners logbook entries, changes in concomitant medications, and adverse events.

The primary objective of the study is to evaluate the efficacy of IGC-AD1 on agitation, measured by changes in the Cohen-Mansfield Agitation Inventory (CMAI) scores from baseline to the End of treatment (EOT). The secondary objective is to assess efficacy by examining CMAI score changes from baseline to week two. Additionally, exploratory objectives are outlined in separate documentation.

Blood samples will be collected during the trial for sparse pharmacokinetic (PK) analysis, blood-based CNS biomarker, and genotyping.

ELIGIBILITY:
To be eligible to participate in this study, the participant must meet all the following criteria:

Inclusion Criteria

1. Participant and/or Caregiver must provide a signed and dated ICF prior to any study procedures.
2. Must have a Caregiver who is able and willing to comply with all required study procedures.
3. The Caregiver must be known to the Participant and must be able to use electronic devices such as a cell phone, video conference over a laptop or cell phone, weighing scale, and be able to learn to take blood pressure, among others.
4. Based on local practice, Participants that cannot consent may have Caregiver's consent provided the Caregiver has among others a) Power of Attorney, b) is a spouse, or c) a sibling or d) a child or e) a close relation. The practice of accepting consent must be consistent with established practice at the site and jurisdiction.
5. Participants must consent to CYP450 and apolipoprotein E (ApoE) genotyping, and pharmacokinetics.
6. Diagnosis of AD by NIA-AA criteria
7. Clinically significant Agitation assessed by:

   1. NPI (Agitation) ≥ 4
   2. The presence of clinically significant, persistent Agitation based on the IPA definition (Appendix C) rather than those with recent onset and occasional symptoms, and
   3. Agitation not attributable to another psychiatric disorder, suboptimal care conditions, other underlining medical condition, or the physiological effects of a substance.
8. Negative drug screen, except for benzodiazepines if Participant has been using them in stable doses for at least 3 months before screening.
9. All medications used for behavioral symptoms should be consistent for at least 6 weeks before screening, with allowance for dose changes up to 25%.
10. Women must be of no childbearing potential (postmenopausal, defined as cessation of menses for at least 12 months, without an alternative medical cause for amenorrhea) or surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation)).

An individual who meets any of the following criteria will be excluded from participation in this study:

Exclusion Criteria

1. Prior adverse reaction to cannabinoids or to any component of Study Drug (IGC-AD1 and placebo).
2. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease, which might confound assessment of safety outcomes.
3. History of seizures, schizophrenia, or bipolar disorder.
4. Has participated in an investigational drug or device study within 30 days prior to study start.
5. Urine drug screen positive for drug use, except for benzodiazepines if Participant was using them previously and their dose had remained stable for at least six weeks before screening.
6. History of Alcohol and Drug use disorder, within one year prior to enrollment.
7. Hypertension: Participants with a history of uncontrolled hypertension as determined by the PI and Participants with a hypertensive crisis in the six months prior to enrollment.
8. Falls: Participants with a history of recurrent falls defined as more than two falls in the six-month period prior to enrollment and a history of falls resulting in injuries or associated with a new acute illness, loss of consciousness, fever, or abnormal blood pressure (Fuller et al., 2000).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Agitation | Baseline to week six
  Change in mean Cohen Mansfield Agitation Inventory (CMAI) score

SECONDARY OUTCOMES:
Acute Agitation | Baseline to week two
  Change in mean Cohen Mansfield Agitation Inventory (CMAI) score

OTHER OUTCOMES:
Agitation at week four | Baseline to week four
  Change in mean Cohen Mansfield Agitation Inventory (CMAI) score
Participant overall wellbeing | Baseline to weeks two and six
  Change in the Clinical Global Impression Scale (CGI)
Participant executive functions | Baseline to week six
  Change in Mini-Mental State Examination (MMSE2) score
Depression | Baseline to weeks two, four, and six
  Change in mean Cornell Scale for Depression in Dementia (CSDD) score
Neuropsychiatric symptoms | Baseline to weeks two, four, and six
  Change in mean Neuropsychiatric Inventory (NPI-12) score
Participant quality of life | Baseline to weeks two, four and six
  Change in mean Quality of Life in Alzheimer's Disease (QOL-AD) score
Caregiver burden | Baseline to weeks two and six
  Change in mean Zarit Burden Interview (ZBI) score
Psychotropic drugs | Baseline to six weeks
  Change in type and dosage of psychotropic drugs
CYP2C9 polymorphisms on agitation | Baseline to weeks two, four and six
  Change in mean Cohen Mansfield Agitation Inventory (CMAI) score for each type of metabolizer group (*1/*1, *1/*3, etc.)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (20):
  - ClinCloud, LLC, Maitland, Florida
  - ClinCloud, LLC, Melbourne, Florida
  - Global Medical Institutes Florida, LLC, Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Miami Jewish Health, Miami, Florida
  - Neurostudies Inc., Port Charlotte, Florida
  - BayCare Health System Inc., St. Petersburg, Florida
  - University of South Florida Department of Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Tandem Intermediate, LLC, Metairie, Louisiana
  - MedStar Franklin Square Medical Center Neurology, Baltimore, Maryland
  - Medstar Georgetown University Hospital Neurology, Clinton, Maryland
  - Medstar Montgomery Medical Center, Olney, Maryland
  - Tekton Research LLC, St Louis, Missouri
  - Dent Neurosciences Research Center, Amherst, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Ichor Research, Syracuse, New York
  - Lynn Health Science Institute (LHSI), Oklahoma City, Oklahoma
  - Butler Hospital, Brown University, Providence, Rhode Island
  - Senior Adults Specialty Research, Austin, Texas
  - Dominion Medical Associates, Inc., Richmond, Virginia
- Canada (4):
  - Island Health Authorities, Victoria, British Columbia
  - Hamilton Health Sciences , Mcmaster University, Hamilton, Ontario
  - Baycrest Academy, University of Toronto, Toronto, Ontario
  - Douglas Hospital Research Center, McGill university, Montreal, Quebec
- Grupo de Neurociencias de Antioquia, Universidad de Antioquia, Medellín, Antioquia, Colombia
- Puerto Rico (3):
  - Instituto Sanacoop, Bayamón, Bayamón
  - SCB Research Center, Bayamón
  - University of Puerto Rico, Rio Piedras

IPD SHARING:
Plan to Share IPD: No